CLINICAL TRIAL: NCT05282433
Title: Surufatinib Alone or Combined With Anti-PD-1 mAb in the Treatment of Advanced Hepatocellular Carcinoma:HCCSC C01 Trial
Brief Title: Surufatinib Alone or Combined With Anti-PD-1 mAb in the Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Clinical Professor of Zhongnan Hospital, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC H01
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; Targeted Therapy; Progression-free Survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Research Group (Experimental): Patients with advanced hepatocellular carcinoma who had failed previous standard 1/2-line therapy and could not tolerate or reject existing therapies.
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib Alone or Combined With Anti-PD-1 mAb in the Treatment of Advanced Hepatocellular Carcinoma
  Other Names: Anti-PD-1 mAb

SUMMARY:
This is an open, prospective, single-arm, multi-cohort clinical study to evaluate the efficacy and safety of surufatinib alone or combined with Anti-PD-1 mAb in the treatment of advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
This is an open, prospective, single-arm, multi-cohort clinical study to evaluate the efficacy and safety of surufatinib alone or combined with Anti-PD-1 mAb in the treatment of advanced Hepatocellular Carcinoma.

Cohort A: patients with advanced hepatocellular carcinoma who had failed previous standard first-line therapy and could not tolerate or reject existing therapies.Treatment:surufatinib combined with Anti-PD-1 mAb Cohort B: patients with advanced pancreatic cancer who had previously failed standard sencond-line therapy, could not tolerate or reject existing therapies.Treatment:surufatinib alone.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years to 75 years. 2.Had a disease status that was measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST, version1.1)： Cohort A: patients with advanced hepatocellular carcinoma who had failed previous standard first-line therapy and could not tolerate or reject existing therapies.

Cohort B: patients with advanced hepatocellular carcinoma who had previously failed standard sencond-line therapy, could not tolerate or reject existing therapies.

3.Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥80g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.5×the upper limit of normal(ULN), ALT and AST≤2.5×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.5 x ULN, creatinine clearance rate > 50ml/min).

4.At least 4 weeks after the last anti-tumor treatment (surgery, chemotherapy, radiotherapy, biotherapy or endocrine therapy) before enrollment.

5.Had a life expectancy of at least 3 months. 6.Had an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2.

7.Signed informed consent.

Exclusion Criteria:

* 1.In the past or at the same time with other malignant tumors (already cure period of IB or cervical, lower levels of noninvasive basal cell or squamous cell cancer, obtain complete remission (CR) > 10 years of breast cancer, obtain complete remission (CR) > 10 years of malignant melanoma, obtain complete remission (CR) > 5 years except of other malignant tumors).

  2.Pregnant or lactating female patients. 3.Had a history of clinically significant or uncontrolled heart disease, including but not limited to: (1)Myocardial infarction. (2)Angina.(3)Congestive heart failure above grade 2 of the New York heart association (NYHA).(4)Ventricular arrhythmias requiring continuous treatment.(5)Supraventricular arrhythmias, including uncontrolled atrial fibrillation.

  4.The patients had mental disorders, and the researchers believed that the patients could not fully or fully understand the possible complications in this study.

  5.Have a history of immunodeficiency, including: HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.

  6.Those who cannot tolerate or may be allergic to the drugs used in this study. 7.Participated in clinical trials of other drugs within the past 1 month. 8.Other factors considered unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-16 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 12 weeks
  Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Fuxiang Zhou, MD,PhD, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China